CLINICAL TRIAL: NCT03269383
Title: Study for the Evaluation of the Effectiveness of Stellate Ganglion Blockade in Preventing Postoperative Atrial Fibrillation
Brief Title: Study to Evaluate the Effectiveness of SGB in Preventing Post-op Atrial Fibrillation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding and other logistical issues
Sponsor: Christopher Connors, MD (Other)
Responsible Party: Sponsor-Investigator, Christopher Connors, MD, Director of Cardiac Anesthesia, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1046118-1
Record Dates: First submitted 2017-06-19; First posted 2017-08-31 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
Keywords: stellate ganglion block; cardiac surgery; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with 2 arms, treatment and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drugs will be randomized and prepared by the institutional pharmacy. The research coordinator will maintain the log tracking which patients received treatment vs placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline (Sham Comparator): Patients will receive a stellate ganglion block but with 10ml of 0.9% saline.
  Interventions: Other: Saline
- Treatment (Experimental): Patients will receive a stellate ganglion block with 10ml of 0.5% bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Patients will receive a stellate ganglion block using 10 ml of 0.5% bupivacaine
  Other Names: marcaine; Sensorcaine
  Arms: Treatment
Other: Saline — Patients will receive a stellate ganglion block using 10 ml of 0.9% saline
  Arms: Saline

SUMMARY:
Atrial fibrillation requires both an initiation trigger and favorable environment for maintenance and the sympathetic and parasympathetic nervous systems play important roles in this regard. Unfortunately, the precise mechanisms of post operative atrial fibrillation (POAF) are still being investigated. This postoperative complication has persisted in spite of efforts to mitigate it pharmacologically with beta blockers and amiodarone, an experience shared by most other cardiac surgery centers.

The stellate ganglion is formed by the fusion of the inferior cervical sympathetic ganglion and first thoracic sympathetic ganglion. By modulating the sympathetic component of the autonomic nervous system, stellate ganglion stimulation has been shown to facilitate induction of atrial fibrillation while ablation may reduce or prevent episodes. Human studies have further supported this model.

Preliminary studies of perioperative stellate ganglion block (SGB) in cardiac surgery suggest that this technique may reduce or prevent episodes of POAF requiring treatment. The investigator's hypothesis is that SGB reduces the incidence of POAF in cardiac surgery populations.

DETAILED DESCRIPTION:
The investigator's hypothesis is that perioperative SGB in cardiac surgery will decrease POAF. To address this, the investigator will:

1. Recruit 707 patients to undergo perioperative SGB prior to cardiac surgery (CABG, Aortic Valve Replacement, CABG/Aortic Valve Replacement).
2. Perform a double blinded post-induction/pre-operative SGB using either 10 mL 0.5% bupivacaine or 10 mL 0.9% normal saline
3. Assess the effects on POAF as defined by the Northern New England (NNE) Cardiovascular Disease Study Group.

Significance: If the investigator is able to demonstrate that perioperative SGB in cardiac surgery affects POAF, this simple, low cost and low risk procedure may significantly impact POAF incidence and thereby its attendant morbidity, mortality and costs in this clinical population.

Study subjects 707 patients electively scheduled for aortic valve, coronary revascularization surgery (CABG) or a combination of the two (CABG/AVR) will be recruited and enrolled to receive SGB at the time of surgery. Patients will be introduced to the study by their surgical team and only those providing informed consent to participate will be enrolled. The informed consent document (attached) clearly states that SGB is not currently standard of care.

Randomization The investigator will use NQuery software (Statistical Solutions Ltd., Boston, MA) to create a randomization scheme stratified by the three types of elective surgery: CABG, aortic valve replacement, and CABG plus aortic valve replacement. Patients will be randomized in a 1:1 ratio to receive either SGB (case, injection of 10 mL 0.5% bupivacaine injection) or sham SGB (control, injection of 10 mL 0.9% saline). For each of the three surgery types, treatment assignments will be placed in opaque envelopes, numbered sequentially; these three series of assignments will be maintained in separate surgery-specific boxes. Medications will be unidentified at the time of injection and the anesthesiologists and cardiac surgeons will be blinded to sham versus treatment group.

Power analysis:

Sample size was calculated based on a group sequential test of two proportions (NQuery, Statistical Solutions Ltd., Boston, MA), which takes into account a single interim analysis of SGB efficacy once 50% of the proposed study group have been enrolled. At 80% power, cumulative alpha = 0.05, with a two-sided test with continuity correction, and using the O'Brien-Fleming spending function, a total study group of n=632 (n=316/ treatment group) would be required to detect a decrease in the rate post-operative atrial fibrillation from 30% to 20% with stellate ganglion block. After taking the interim analysis (performed when n=350; significance accepted at p<0.003) into account, significance will be accepted at p<0.047 for the overall study. In our preliminary feasibility study, the investigator established that stellate ganglion block was successful in 88% of cases; thus, the sample size was increased by 12%, from n=632 to n=707.

Data analysis. Descriptive statistics (mean (SD), median, frequency as appropriate) will be used to summarize the demographic, procedural and clinical characteristics of the study group. To evaluate the success of randomization, the investigator will describe demographic and clinical data both overall and after stratification by surgery type and by treatment type. As intra-operative conditions can direct modification in the actual surgery performed (e.g. CABG may become CABG plus valve replacement), the investigator will also describe the proportion of subjects who were misclassified by surgery type during randomization and if necessary will assess randomization balance according to the actual surgery type received.

The frequency of atrial fibrillation (AF) will be compared between treatment groups by chi square test; this primary analysis will be performed first using an intention to treat model. In post hoc analysis the investigator will explore treatment outcomes after stratification by type of surgery and established clinical risk factors for POAF (age, sex, smoking, obesity, hypertension, diabetes mellitus, myocardial infarction, and BMI). If descriptive analyses suggest imbalance in clinical or demographic characteristics between treatment groups, these will be explored using t tests or their non-parametric equivalent (continuous data) or chi square test (categorical data), as appropriate, and logistic regression will be used to evaluate differences in AF rate between treatment groups, while taking identified covariates into account.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for non-emergent CABG, AVR, or CABG/AVR
* aged at least 18 years
* English speaking

Exclusion Criteria:

* aged less than 18 years
* pregnant women
* prisoners
* patients having emergency surgery
* patients with clinical contraindications to SGB (including allergy to local anesthetic, carotid vascular disease as defined by ipsilateral prior carotid endarterectomy or carotid stent, superficial infection at the proposed puncture site, contralateral phrenic or laryngeal nerve palsies, and severe chronic obstructive pulmonary disease as defined by the need for home oxygen)
* patients who are unable to provide informed consent for themselves
* patients with a history of atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation | up to 7 days
  looking for absence of new onset postoperative atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Chris Connors, MD, Principal Investigator — Spectrum Medical Group, Maine Medical Center
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mostafa A, El-Haddad MA, Shenoy M, Tuliani T. Atrial fibrillation post cardiac bypass surgery. Avicenna J Med. 2012 Jul;2(3):65-70. doi: 10.4103/2231-0770.102280. PMID 23826549
- [Background] Zhou Q, Hu J, Guo Y, Zhang F, Yang X, Zhang L, Xu X, Wang L, Wang H, Hou Y. Effect of the stellate ganglion on atrial fibrillation and atrial electrophysiological properties and its left-right asymmetry in a canine model. Exp Clin Cardiol. 2013 Winter;18(1):38-42. PMID 24294036
- [Background] Al-Atassi T, Toeg H, Malas T, Lam BK. Mapping and ablation of autonomic ganglia in prevention of postoperative atrial fibrillation in coronary surgery: MAAPPAFS atrial fibrillation randomized controlled pilot study. Can J Cardiol. 2014 Oct;30(10):1202-7. doi: 10.1016/j.cjca.2014.04.018. Epub 2014 Apr 19. PMID 25262862
- [Background] Yildirim V, Akay HT, Bingol H, Bolcal C, Iyem H, Doganci S, Demirkilic U, Tatar H. Pre-emptive stellate ganglion block increases the patency of radial artery grafts in coronary artery bypass surgery. Acta Anaesthesiol Scand. 2007 Apr;51(4):434-40. doi: 10.1111/j.1399-6576.2006.01260.x. PMID 17378781
- [Background] Bidwai AV, Rogers CR, Pearce M, Stanley TH. Preoperative stellate-ganglion blockade to prevent hypertension following coronary-artery operations. Anesthesiology. 1979 Oct;51(4):345-7. doi: 10.1097/00000542-197910000-00015. No abstract available. PMID 314762
- [Background] Donmez A, Tufan H, Tutar N, Araz C, Sezgin A, Karadeli E, Torgay A. In vivo and in vitro effects of stellate ganglion blockade on radial and internal mammary arteries. J Cardiothorac Vasc Anesth. 2005 Dec;19(6):729-33. doi: 10.1053/j.jvca.2004.10.008. PMID 16326296
- [Background] Garneau SY, Deschamps A, Couture P, Levesque S, Babin D, Lambert J, Tardif JC, Perrault LP, Denault AY. Preliminary experience in the use of preoperative echo-guided left stellate ganglion block in patients undergoing cardiac surgery. J Cardiothorac Vasc Anesth. 2011 Feb;25(1):78-84. doi: 10.1053/j.jvca.2010.03.007. Epub 2010 Jun 30. PMID 20580574
- [Background] Gopal D, Singh NG, Jagadeesh AM, Ture A, Thimmarayappa A. Comparison of left internal mammary artery diameter before and after left stellate ganglion block. Ann Card Anaesth. 2013 Oct-Dec;16(4):238-42. doi: 10.4103/0971-9784.119161. PMID 24107689
- [Background] Haest K, Kumar A, Van Calster B, Leunen K, Smeets A, Amant F, Berteloot P, Wildiers H, Paridaens R, Van Limbergen E, Weltens C, Janssen H, Peeters S, Menten J, Vergote I, Morlion B, Verhaeghe J, Christiaens MR, Neven P. Stellate ganglion block for the management of hot flashes and sleep disturbances in breast cancer survivors: an uncontrolled experimental study with 24 weeks of follow-up. Ann Oncol. 2012 Jun;23(6):1449-54. doi: 10.1093/annonc/mdr478. Epub 2011 Oct 29. PMID 22039079
- [Background] Kumar N, Thapa D, Gombar S, Ahuja V, Gupta R. Analgesic efficacy of pre-operative stellate ganglion block on postoperative pain relief: a randomised controlled trial. Anaesthesia. 2014 Sep;69(9):954-660. doi: 10.1111/anae.12774. Epub 2014 Jul 7. PMID 25040168
- [Background] Wulf H, Maier C. [Complications and side effects of stellate ganglion blockade. Results of a questionnaire survey]. Anaesthesist. 1992 Mar;41(3):146-51. German. PMID 1570888
- [Background] Stoller JK, Panos RJ, Krachman S, Doherty DE, Make B; Long-term Oxygen Treatment Trial Research Group. Oxygen therapy for patients with COPD: current evidence and the long-term oxygen treatment trial. Chest. 2010 Jul;138(1):179-87. doi: 10.1378/chest.09-2555. PMID 20605816